CLINICAL TRIAL: NCT05988905
Title: The Effects of Gait Performance and Brain Activity After Robot-assisted Gait Training (RAGT) On Patients With Lower Extremity Thermal Injury : a Prospective, Randomized, Single-blinded Study
Brief Title: The Effects of Gait Performance and Brain Activity After Robot-assisted Gait Training (RAGT) On Patients With Lower Extremity Thermal Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hangang Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, So Young Joo, Hangang Sacred Heart Hospital, Hangang Sacred Heart Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HangangSHH-17
Record Dates: First submitted 2023-08-03; First posted 2023-08-14 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Gait Disorder, Sensorimotor
Keywords: robot; burn patient; functional near-infrared spectroscopy
MeSH Terms: conditions — Gait Disorders, Neurologic

STUDY DESIGN:
Intervention Model Description: robot assisted gait training
Who Masked: Outcomes Assessor
Masking Description: Robot assisted gait training enables training of automatically programmed normal gait pattern. Patients underwent 30 min of RAGT using SUBAR® and conventional exercise rehabilitation each for 30 min once a day for 5 days a week for 8 weeks. The CON group focused on gait training such as active range of motion (ROM) exercise, weight bearing training, manual lymphatic drainage, and hypertrophic scar care for 60 min once a day for 5 days a week for 8 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- robot assisted gait training (Experimental): RAGT enables training of automatically programmed normal gait pattern. Patients underwent 30 min of RAGT using SUBAR® and conventional exercise rehabilitation each for 30 min once a day for 5 days a week for 8 weeks.
  Interventions: Other: robot assited gati training
- conventioanl training (Active Comparator): The conventional training group focused on gait training such as active range of motion (ROM) exercise, weight bearing training, manual lymphatic drainage, and hypertrophic scar care for 60 min once a day for 5 days a week for 8 weeks.
  Interventions: Other: conventional traiing

INTERVENTIONS:
Other: robot assited gati training — SUBAR® (CRETEM, Korea) is a exoskeletal-robot with a footplate that assists gait movements. The patient's thigh length and lower leg length were measured before training, so that the SUBAR® can be adjusted to patient's size to ensure accurate training. During training, the therapist facilitated the treatment and stood by the patients' side to adjust the direction and speed. RAGT is programmed automatically, and it can be performed regularly over a long period. The patients received 30 min of robot-assisted training using SUBAR® once a day for 5 days a week for 8 weeks. Each training session lasted up to 40 min.
  Arms: robot assisted gait training
Other: conventional traiing — Patients also received conventional exercise rehabilitation with the same duration and frequency. Conventional rehabilitation therapy, which consisted of active assistive knee exercises, knee stretching, patellar mobilization exercises, and quadriceps setting exercises, was performed every day throughout the rehabilitation period.
  Arms: conventioanl training

SUMMARY:
Gait enables individuals to move forward and is considered a natural skill. Gait disturbances are very common in patients with burn injury. Major causes of gait disturbances are pain and joint contractures. Recent studies focused on the application of robot-assisted gait training (RAGT) for improving gait functions. This study aimed to elucidate the efficacy and investigate the mechanism of motor recovery after RAGT on patients with lower extremity burn. To investigate the clinical effects, the investigators compare the results of RAGT group to the results of matched conventional (CON) rehabilitation group.This single-blinded, randomized, controlled trial involved 40 patients with lower extremity burns. Patients were randomized into a RAGT or a CON group. SUBAR® (CRETEM, Korea) is a exoskeletal-robot with a footplate that assists patients to perform gait motions. RAGT enables training of automatically programmed normal gait pattern. Patients underwent 30 min of RAGT using SUBAR® and conventional exercise rehabilitation each for 30 min once a day for 5 days a week for 8 weeks. The CON group focused on gait training such as active range of motion (ROM) exercise, weight bearing training, manual lymphatic drainage, and hypertrophic scar care for 60 min once a day for 5 days a week for 8 weeks.A wearable functional near-infrared spectroscopy (fNIRS) device has been developed for studying cortical hemodynamics. Changes in cortical activity has not previously been documented in patients with burn injury. The primary outcome was the prefrontal cortical activity in the both groups. The walking-related cortical activity using an fNIRS device before and after 8 weeks training were measured. To evaluate functional recovery, functional ambulation category (FAC) scores and 6-minute walking test (6MWT) distances were measured. Numeric rating scale (NRS) was used to rate the degree of subjective pain during gait movement: 0 points were assigned when no pain was noted, and unbearable pain was assigned 10 points.

DETAILED DESCRIPTION:
Gait enables individuals to move forward and is considered a natural skill. Gait disturbances are very common in patients with burn injury. Major causes of gait disturbances are pain and joint contractures. Recent studies focused on the application of robot-assisted gait training (RAGT) for improving gait functions. This study aimed to elucidate the efficacy and investigate the mechanism of motor recovery after RAGT on patients with lower extremity burn. To investigate the clinical effects, the investigators compare the results of RAGT group to the results of matched conventional (CON) rehabilitation group.This single-blinded, randomized, controlled trial involved 40 patients with lower extremity burns. Patients were randomized into a RAGT or a CON group. SUBAR® (CRETEM, Korea) is a exoskeletal-robot with a footplate that assists patients to perform gait motions. RAGT enables training of automatically programmed normal gait pattern. Patients underwent 30 min of RAGT using SUBAR® and conventional exercise rehabilitation each for 30 min once a day for 5 days a week for 8 weeks. The CON group focused on gait training such as active range of motion (ROM) exercise, weight bearing training, manual lymphatic drainage, and hypertrophic scar care for 60 min once a day for 5 days a week for 8 weeks.A wearable functional near-infrared spectroscopy (fNIRS) device has been developed for studying cortical hemodynamics. Changes in cortical activity has not previously been documented in patients with burn injury. The primary outcome was the prefrontal cortical activity in the both groups. The walking-related cortical activity using an fNIRS device before and after 8 weeks training were measured. To evaluate functional recovery, functional ambulation category (FAC) scores and 6-minute walking test (6MWT) distances were measured. Numeric rating scale (NRS) was used to rate the degree of subjective pain during gait movement: 0 points were assigned when no pain was noted, and unbearable pain was assigned 10 points.

ELIGIBILITY:
Inclusion Criteria:

* patients with full or virtually full thickness involvement of >50% on the body surface area of the bilateral lower extremity
* age > 18 years
* with ≤1 functional ambulation category (FAC) score ≤ 3

Exclusion Criteria:

* patients with cognitive disorders
* intellectual impairment before burn injury
* serious cardiac dysfunction
* problems with weight bearing due to unstable fractures
* body weight ≥100 kg
* severe fixed contracture
* skin disorders that could be worsened by RAGT and conventional rehabilitation
* patients with severe pain who were unable to undergo conventional rehabilitation programs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
near infrared spectroscopy | 8 weeks
  The rest period before gait period served as a baseline reference for osyhemoglobin of PFC perfusion. Cortical activity was measured by evaluating relative changes in oxyhemoglobin level and deoxyhemoglobin level.

SECONDARY OUTCOMES:
numeric rating scale (NRS) | 8 weeks
  rate the degree of subjective pain during gait movement: 0 points were assigned when no pain was noted, and unbearable pain was assigned 10 points.
functional ambulatory category | 8 weeks
  FAC was evaluated based on six scales. Scale 0 means that the patient cannot walk or can only walk with assistance of two people. Scale 5 means that the patient can walk independently.
6 minutes walking test | 8 weeks
  Patients were instructed to walk as far as possible in 6 min

CONTACTS AND LOCATIONS:
Overall Officials: SO YOUNG JOO, MD, Principal Investigator — handgang sacred heart hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Knaepen K, Mierau A, Swinnen E, Fernandez Tellez H, Michielsen M, Kerckhofs E, Lefeber D, Meeusen R. Human-Robot Interaction: Does Robotic Guidance Force Affect Gait-Related Brain Dynamics during Robot-Assisted Treadmill Walking? PLoS One. 2015 Oct 20;10(10):e0140626. doi: 10.1371/journal.pone.0140626. eCollection 2015. PMID 26485148
- [Result] Hawkins KA, Fox EJ, Daly JJ, Rose DK, Christou EA, McGuirk TE, Otzel DM, Butera KA, Chatterjee SA, Clark DJ. Prefrontal over-activation during walking in people with mobility deficits: Interpretation and functional implications. Hum Mov Sci. 2018 Jun;59:46-55. doi: 10.1016/j.humov.2018.03.010. Epub 2018 Mar 29. PMID 29604488